CLINICAL TRIAL: NCT03089515
Title: Small Airway Chronic Obstructive Disease Syndrome Following Exposure to WTC Dust
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-01589
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Lower Respiratory Disease
Keywords: World Trade Center; World Trade Center Survivors
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: * Healthy Controls who were not in the WTC program (n = 20)
  * Uncontrolled Lower Respiratory Symptoms in WTC Surivivors; ULRS study) with persistent LRS (n = 40)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Controls (Active Comparator)
  Interventions: Other: Cardio-Pulmonary Exercise Testing (CPET)
- Survivors (Experimental)
  Interventions: Other: Cardio-Pulmonary Exercise Testing (CPET)

INTERVENTIONS:
Other: Cardio-Pulmonary Exercise Testing (CPET) — This test helps determine if the decreased tolerance to exercise or shortness of breath with activity a patient is experiencing is caused by a cardiac disease, versus a pulmonary disease.

SUMMARY:
Many "Survivors" in the World Trade Center (WTC) clinical program have a clinical syndrome characterized by chronic obstruction in small airways and persistence of lower respiratory symptoms despite therapy. This study will test the hypothesis that persistent symptoms in WTC "Survivors" are associated with abnormal small airways whose dysfunction is amplified during exercise and is associated with biologic evidence of inflammation and remodeling. The results from this study will have important treatment implications for our WTC population with potential applicability to larger populations with either inhalational lung injury and/or airway diseases such as asthma and chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

sACOS patients

* Previously participated in ULRS study and signed consent to be recontacted, or
* Patient in the WTC EHC and signed consent to be recontacted
* Onset of lower respiratory symptoms (LRS) after 9/11/01
* ACT < 20 at WTC EHC Monitoring visit
* Presence of LRS on Study Visit 1
* ACT<20 at Study Visit 1
* FEV1 > 70% predicted Study Visit 1
* Using ICS/LABA (Advair HFA equivalent > 115/21 mcg bid) or Fluticasone (110 mcg bid or equivalent) for at least 1 month before Study Visit 1
* CXR without parenchymal abnormalities

Control

* Patient in the WTC EHC and signed consent to be recontacted
* of lower respiratory symptoms on WTC EHC Monitoring Visit of WTC EHC
* Absence of lower respiratory symptoms on Study Visit 1
* FEV1 > 70% predicted on monitoring
* Not on any ICS/LABA/LAMA

Exclusion Criteria:

sACOS

* >10py tobacco use
* Unstable cardiac disease
* Systolic BP > 180 mmHg or Diastolic BP > 120 mmHg
* Oxygen saturation < 90%
* Uncontrolled HTN, DM
* Musculoskeletal inability to exercise
* Use of long acting muscarinic antagonist in the past 2 weeks
* Current use of oral corticosteroids
* Other pulmonary disease, including sarcoidosis, ILD
* Currently pregnant or with plans to become pregnant or lactating
* History of narrow angle glaucoma
* Known prostate hyperplasia or bladder-neck obstruction

Control

* >10py tobacco use
* Unstable cardiac disease
* Systolic BP > 180 mmHg or Diastolic BP > 120 mmHg
* Oxygen saturation < 90%
* Uncontrolled HTN, DM
* Musculoskeletal inability to exercise
* Use of ICS/LABA/SABA/LAMA individually or in combined formulation
* Current use of oral corticosteroids
* Other pulmonary disease, including sarcoidosis, ILD
* Currently pregnant or with plans to become pregnant or lactating
* History of narrow angle glaucoma
* Known prostate hyperplasia or bladder-neck obstruction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Resting Lung Function using Spirometry following Forced Oscillation Techniques | 4 Months
  functional impairment at rest and with increased respiratory frequency (spirometry and forced oscillation techniques; FOT).
Measure of Lung Function using spirometry after inhalation of a targeted anti-muscarinic agent. | 4 Months
  Spirometry (meaning the measuring of breath) is the most common of the pulmonary function tests (PFTs), measuring lung function, specifically the amount (volume) and/or speed (flow) of air that can be inhaled and exhaled.

SECONDARY OUTCOMES:
Comparison of measure of serum marker IL-6 | 4 Months
  Inflammation is caused by extra protein released from the site of inflammation that circulates in the bloodstream. The erythrocyte sedimentation rate (ESR), C-reactive protein (CRP) and plasma viscosity (PV) blood tests are commonly used to detect this increase in protein. In this way they are used as markers of inflammation.
Comparison of measure of serum marker IL-8 | 4 Months
  Inflammation is caused by extra protein released from the site of inflammation that circulates in the bloodstream. The erythrocyte sedimentation rate (ESR), C-reactive protein (CRP) and plasma viscosity (PV) blood tests are commonly used to detect this increase in protein. In this way they are used as markers of inflammation.
Comparison of measure of serum marker CRP | 4 Months
  Inflammation is caused by extra protein released from the site of inflammation that circulates in the bloodstream. The erythrocyte sedimentation rate (ESR), C-reactive protein (CRP) and plasma viscosity (PV) blood tests are commonly used to detect this increase in protein. In this way they are used as markers of inflammation.
Th2 inflammation By measure of fibrinogen | 4 Months
  Inflammation is caused by extra protein released from the site of inflammation that circulates in the bloodstream. The erythrocyte sedimentation rate (ESR), C-reactive protein (CRP) and plasma viscosity (PV) blood tests are commonly used to detect this increase in protein. In this way they are used as markers of inflammation.
Th2 inflammation By measure of periostin | 4 Months
  Inflammation is caused by extra protein released from the site of inflammation that circulates in the bloodstream. The erythrocyte sedimentation rate (ESR), C-reactive protein (CRP) and plasma viscosity (PV) blood tests are commonly used to detect this increase in protein. In this way they are used as markers of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Berger, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States